CLINICAL TRIAL: NCT02183480
Title: Assessment of Dose Proportionality of Different Dose Strengths of Linagliptin Tablets After Oral Administration to Healthy Male and Female Volunteers in an Open, Randomised, Multiple-dose, Three-period Crossover, Phase I Trial
Brief Title: Dose Proportionality of Different Dose Strengths of Linagliptin Tablets After Oral Administration to Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1218.33
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin

ARMS (3):
- Linagliptin, low dose (Experimental)
  Interventions: Drug: Linagliptin, low dose
- Linagliptin, medium dose (Experimental)
  Interventions: Drug: Linagliptin, medium dose
- Linagliptin, high dose (Active Comparator)
  Interventions: Drug: Linagliptin, high dose

INTERVENTIONS:
Drug: Linagliptin, low dose
  Arms: Linagliptin, low dose
Drug: Linagliptin, medium dose
  Arms: Linagliptin, medium dose
Drug: Linagliptin, high dose
  Arms: Linagliptin, high dose

SUMMARY:
Study to assess the pharmacokinetics and dose proportionality of 1 mg, 2.5 mg and 5 mg tablets of linagliptin

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead ECG (electrocardiogram), clinical laboratory tests
* Age 18 to 55 years (inclusive)
* BMI (Body Mass Index) 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance. Repeated measurement of a systolic blood pressure greater than 140 mmHg or diastolic blood pressure greater than 90 mmHg
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs within one month or less than 10 half-lives of the respective drug prior to first study drug administration except if a relevant interaction can be ruled out
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Alcohol abuse ( average consumption of more than 20 g/day in females and 30 g/day in males)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site

For female subjects only:

* Positive pregnancy test, pregnancy or planning to become pregnant during the study or within 2 months after study completion
* No adequate contraception during the study and until 1 month after study completion, i.e. not any of the following: implants, injectables, combined oral contraceptives, IUD (intrauterine device), sexual abstinence for at least 1 month prior to enrolment, vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (including hysterectomy). Females, who do not have a vasectomised partner, are not sexually abstinent or surgically sterile will be asked to use an additional barrier method (e.g. condom, diaphragm with spermicide)
* Lactation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) of linagliptin | up to 168 hours after first drug administration at each visit
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) of linagliptin | up to 168 hours after first drug administration at each visit
Cτ,ss (average measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) of linagliptin | up to 168 hours after first drug administration at each visit

SECONDARY OUTCOMES:
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) of CD 1750 | up to 168 hours after first drug administration at each visit
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) of CD 1750 | up to 168 hours after first drug administration at each visit
Number of patients with adverse events | up to 53 days
Assessment of tolerability by investigator on a 4-point scale | within 10 days after last study drug administration